CLINICAL TRIAL: NCT06294535
Title: The Accuracy of Reconstruction of Orbital Walls Fracture Using Prebent Mesh Versus Patient Specific Implant : A Prospective Study
Brief Title: The Accuracy of Reconstruction of Orbital Walls Fracture Using Prebent Mesh Versus Patient Specific Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, mona samy sheta, lecturer of oral and maxillofacial surgery department, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Orbital Fractures
Keywords: orbital wall reconstruction; prebent titanium mesh; patient specific implant; PEEK
MeSH Terms: conditions — Orbital Fractures

STUDY DESIGN:
Who Masked: Participant
Masking Description: patient select randomly from closed label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prebent titanium mesh (Experimental): reconstruction of fractured orbital walls with perbent titanium mesh
  Interventions: Device: reconstruction of orbital walls
- customized titanium implant (patient specific implant) (Experimental): econstruction of fractured orbital walls with patient specific implant (customized titanium implant)
  Interventions: Device: reconstruction of orbital walls

INTERVENTIONS:
Device: reconstruction of orbital walls — under GA, incision to access to orbital walls. Then insertion of prebent titanium mesh or customized titanium implant and fixation with miniscrews, examination of ocular motility using forced duction test followed by closure of flap.

SUMMARY:
under GA, incision to access to orbital walls. Then insertion of prebent titanium mesh or customized titanium implant and fixation with miniscrews, examination of ocular motility using forced duction test followed by closure of flap.

DETAILED DESCRIPTION:
under GA, incision to access to orbital walls. complete reflection of orbital floor to be constructed then insertion of customized orbital implant of patient or insertion of titanium mrsh after adaption on the model and fixation with miniscrews, examination of ocular motility using forced duction test followed by closure of flap.

ELIGIBILITY:
Inclusion Criteria:

* patient had fractured orbital walls suffering from enophthalmous, hypoglobus, diplopia

Exclusion Criteria:

* systemic disease interfere with bone healing enophthamous less than 2 mm

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
restoring the accurate position of eye | one month- six months
  using exophthalmometer to measure enophthalmous
motility of eye | one month
  using 9 gaze test to evaluate motility of eye
volume of orbit | one to six months
  using CT scan to measure orbital volume pre and postoperative

CONTACTS AND LOCATIONS:
Overall Officials: mona s sheta, lecturer, Principal Investigator — Tanta University
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt